CLINICAL TRIAL: NCT03498157
Title: IMpact of PRehabilitation in Oncology Via Exercise - Breast Cancer
Acronym: IMPROVE-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Kathryn Schmitz, Professor, Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PSCI # 17-051
Record Dates: First submitted 2018-02-21; First posted 2018-04-13 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer; Prehabilitation; Physical Activity; Surgery
Keywords: Prehabilitation; Exercise; Breast Cancer; Physical Activity; Surgery
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Partly Supervised Prehabilitation (Experimental): Will be offered an initial one week (5 days for 3 hours each) supervised exercise prehabilitation program including a two hour group-based prehabilitation class at Penn State Rehabilitation Hospital, Hummelstown. The following weeks till surgery the learned exercise program should be done home-based for 5 times a week. A weekly phone call during this period will help to support and adapt the exercise program.
  Interventions: Behavioral: Exercise; Behavioral: Prehabilitation Education
- Home-based Prehabilitation (Active Comparator): Will be offered an individual one-on-one appointment for an exercise introduction session with an exercise and cancer specialist and weekly phone calls to support and adapt the exercise program. The exercises should be done home-based for 5 times a week until the time of surgery. Furthermore, a two hour group-based prehabilitation class at the Penn State Hershey Cancer Institute will be offered.
  Interventions: Behavioral: Exercise; Behavioral: Prehabilitation Education
- Control Group (Active Comparator): Will be offered a two hour group-based prehabilitation class at the Penn State Hershey Cancer Institute.
  Interventions: Behavioral: Prehabilitation Education
- Comparison group- women too active (No Intervention): Added comparison group: Women who are ineligible on the basis of 'engaging in systematic intense exercise training (at least 1h twice a week) will be recruited to complete measures only, with no randomization

INTERVENTIONS:
Behavioral: Exercise — The exercise intervention is an at least 2 weeks lasting (till the day surgery is taking place) 5-times weekly resistance training intervention combined with aerobic exercise (mostly walking).
  Arms: Home-based Prehabilitation; Partly Supervised Prehabilitation
Behavioral: Prehabilitation Education — Participate will receive a 2 hour group-based prehabilitation class which will be held at the Penn State Cancer Institute, Hershey
  Arms: Control Group; Home-based Prehabilitation; Partly Supervised Prehabilitation

SUMMARY:
The purpose of this study is to determine whether patients are able to participate in a so called prehabilitation program (prior to the beginning of cancer treatment) which includes (1) a supervised and home-based exercise program plus one educational session or (2) just home-based exercise plus one educational session or (3) just one educational session.

Breast cancer surgery may have potential for several side effects, including functional (e.g. flexibility in the affected arm, lymphedema [swelling that generally occurs in the arms or legs that occurs as a result of the removal of or damage to lymph nodes as a part of cancer treatment], shoulder pain) and psychosocial (e.g. reduced quality of life, increased fatigue) aspects.

Evidence shows that exercise is considered to be an effective treatment approach in breast cancer patients during and after treatment with regard to the above mentioned side-effects. Also, prehabilitative exercise in colon and lung cancer patients was shown as feasible and effective. However, no experience exits with regard to prehabilitation exercise in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral primary carcinoma of the breast, confirmed histologically by core biopsy
* Not metastatic (stage <4)
* Females and males ≥18 years of age
* Fluent in written and spoken English
* Must be able to provide and understand informed consent
* Must have an ECOG PS of ≤ 2
* Scheduled for lump- or mastectomy at Penn State Cancer Institute
* ≥ 2 weeks till primary treatment
* Primary attending surgeon approval

Exclusion Criteria:

* Receiving neoadjuvant chemotherapy, radiotherapy or hormone therapy
* Not fluent in written and spoken English
* Evidence in the medical record of an absolute contraindication (e.g. Heart insufficiency > NYHA III or uncertain arrhythmia; uncontrolled hypertension; severe renal dysfunction (GFR < 30%, Creatinine> 3mg/dl; insufficient hematological capacity like either hemoglobin value below 8 g/dl or thrombocytes below 30.000/µL; reduced standing or walking ability) for exercise
* Pregnant women
* Engaging in systematic intense exercise training (at least 1h twice per week)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Safety of the exercise intervention (assessed by standardized questionnaire) | Through study intervention, an average of 3 weeks
  Within the questionnaire we will assess whether musculoskeletal occur (yes/no; ongoing; location; severity (mild-life threatening); daily activities affected). The intervention will be considered as safe if less than 25% of included patients report mild musculoskeletal impairments and less than 5% experienced musculoskeletal injuries (defined as symptoms lasting a week or longer and or requiring the attention of a medical professional).
Feasibility of the exercise intervention (assessed via exercise logs) | Through study intervention, an average of 3 weeks
  The exercise intervention will be considered feasible if 50% of included patients actually do at least half of the exercise sessions prescribed for 2 weeks or more.
Acceptability of the exercise intervention (assessed via patient flow diagram) | During Recruitment till first intervention is delivered (with one week after enrolment)
  The intervention will be considered acceptable if more than 50% of the patients randomized to the control group agree to receive at least the first exercise session.

SECONDARY OUTCOMES:
Health-Related Quality of Life: EORTC QLQ-C30, version 3.0 | Through study intervention, an average of 3 weeks; 6 weeks after surgery; and after the end of primary treatment, an average of 6 month after surgery
  QoL will be assessed with the validated 30-item self-assessment questionnaire of the European Organization for Research and Treatment of Cancer (EORTC QLQ-C30, version 3.0).
Breast cancer-related symptoms and quality of Life | Through study intervention, an average of 3 weeks; 6 weeks after surgery; and after the end of primary treatment, an average of 6 month after surgery
  In addition to the EORTC-QLQ-C30 specific breast cancer-related symptoms will be assessed with the validated 23-item breast cancer specific module (EORTC QLQ-BR23). It will assess common problems of breast cancer patients, e.g. with the affected breast or arm
Fatigue | Through study intervention, an average of 3 weeks; 6 weeks after surgery; and after the end of primary treatment, an average of 6 month after surgery
  Fatigue will be assessed with the Multidimensional Fatigue Inventory (MFI) which is a 20-item, multidimensional self-assessment questionnaire.
Sleep | Through study intervention, an average of 3 weeks; 6 weeks after surgery; and after the end of primary treatment, an average of 6 month after surgery
  Sleep quality and sleep problems will be assessed with the validated and frequently used Pittsburgh Sleep Quality Index (PSQI)
Depression | Through study intervention, an average of 3 weeks; 6 weeks after surgery; and after the end of primary treatment, an average of 6 month after surgery
  Depressive symptoms will be assessed with the 20-item Center for Epidemiological Studies Depression Scale (CES-D).
Shoulder Problems | Through study intervention, an average of 3 weeks; 6 weeks after surgery; and after the end of primary treatment, an average of 6 month after surgery
  The Penn Shoulder Score (PSS) is a 100-point shoulder-specific self-report questionnaire consisting of 3 subscales of pain, satisfaction, and function.
Physical activity behavior | Through study intervention, an average of 3 weeks; 6 weeks after surgery; and after the end of primary treatment, an average of 6 month after surgery
  Physical activity behavior in the domains of commuting activity, leisure time activities such as cycling, walking, and sports, household and occupational activity will be assessed via a standardized and validated questionnaire, the Short QUestionnaire to ASsess Health-enhancing Physical Activity
Symptoms | Weekly from baseline to 6 weeks after Surgery
  The revised Edmonton symptom assessment scale is a 10-item patient-rated symptom visual numeric scale developed for use in assessing symptoms of patients receiving palliative care/cancer treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M Schmitz, PhD, Principal Investigator — Penn State College of Medicine Hershey; Joachim Wiskemann, PhD, Principal Investigator — National Center for Tumor Diseases, Heidelberg
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No